CLINICAL TRIAL: NCT06566677
Title: Validation of Selected Point of Care Rapid STI Diagnostic Tests for Laboratory Based and Self- Test Use - A Sub-Study of Acceptability Research on Integrated Point of Care Sexually Transmitted Infection (STI) Testing and Expanded Partner Therapy (EPT) (ARISE)
Brief Title: Point of Care Rapid STI Test Optimization and Validation Extension
Acronym: PROVE
Status: Completed | Type: Observational
Sponsor: Wits RHI Research Centre Clinical Research Site (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Thesla Palanee-Phillips, Director of Clinical Trials, Wits RHI Research Centre Clinical Research Site
Other Study IDs: PROVE
Record Dates: First submitted 2024-08-16; First posted 2024-08-22 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Chlamydia Trachomatis Genital Infection; Gonorrhea; Trichomoniasis
MeSH Terms: conditions — Gonorrhea; Trichomonas Infections

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biological specimens such as blood and vaginal fluid will be used to validate commercially available point of care diagnostic STI tests for Neisseria gonorrhoea (NG), Chlamydia trachomatis (CT) and Trichomonas vaginalis (TV) as well as other STIs where applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this sub-study (PROVE) is to support and facilitate the validation of commercially available point of care (POC) sexually transmitted infection (STI) diagnostic test kits/devices for potential on-site laboratory use as well as bedside use in parallel to gold standard established testing methodologies. A further extension of bedside testing would include self-testing.

DETAILED DESCRIPTION:
Screening and Enrolment procedures for the ARISE study (HREC Ref No. 210614) involves adolescent girls and young women (AGYW) being screened for Neisseria gonorrhoea (NG), Chlamydia trachomatis (CT), and Trichomonas vaginalis (TV) as determined through testing of clinician-collected genital swabs followed by GeneXpert, OSOM rapid TV testing or through wet mount visualisation of the micro-organisms of interest. This will generate a pool of AGYW with known STI diagnoses who, if positive, will be treated on-site on the day of STI detection. It will also create an ideal opportunity to leverage access to samples from willing participants (prior to STI treatment if STI positive) for validation of a range of alternate STI test kits. Samples provided will enable same-day parallel testing on additional platforms for validation of the sensitivity and specificity of these alternate tests against the known validated platformsThis initiative will expand the menu of cost effective and user friendly STI test kits that may ultimately be used in other research studies, in public clinic settings and as self-tests performed discretely in the convenience and privacy of one's home.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria to be eligible for inclusion in the study:

* Cisgender adolescent girls and young women (18-25 years of age, inclusive), screened for or enrolled in the ARISE study.
* Willing to provide written informed consent to participate in this sub-study.
* Willing to provide additional samples including vaginal and endocervical swabs, urine and those collected through the use of tampons and disposable menstrual cups.

Exclusion Criteria:

* Cisgender male or transgender woman or transgender man
* Age <18 years
* Unable or unwilling to provide written informed consent
* Have any condition that in the opinion of the investigators will interfere with successful completion of sub-study procedures

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender females.
Study Population: Participants screened and/or enrolled into ARISE (HREC Ref No. 210614): Sexually active non-pregnant, HIV-negative, cis-gender AGYW aged 18-25
Sampling Method: Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
GeneXpert | 1 year
  A PCR instrument was used to assess the presence of chlamydia trichomatis and gonorrhea from samples taken using endocervical swabs.

SECONDARY OUTCOMES:
Osom rapid testing kit | 1 year
  A rapid point-of-care test for the diagnosis of Trichomonas vaginalis in women using dacron swabs.

OTHER OUTCOMES:
JD Biotech Trichomonas vaginalis antigen rapid test kit | 1 year
  Trichomonas vaginalis antigen rapid test kit
JD Biotech C. Trachomatis/ N. Gonorrhoeae Ag combo rapid test | 1 year
  Urine or vaginal cavity swab or vaginal glans sample to diagnose chlamydia trichomati and gonorroea
Cromatest Chlamydia one step rapid kit | 1 year
  Female cervical swab and male urethral swab specimens to diagnose chlamydia
NADAL Chlamydia Test | 1 year
  Female or male urethral swab/male Urine used to diagnose chlamydia
ACRO Biotech Gonorrhoea | 1 year
  Female cervical swab/ male urethral swab to diagnose gonorrhoea
Rapid Labs Gonorrhea | 1 year
  Sterile Female cervical swab/ male urethral swab to diagnose gonorrhea

CONTACTS AND LOCATIONS:
Locations (1):
- Wits RHI Research Centre, Hillbrow, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No
Results of the validations will be shared with study staff, study participants, CAB members and other key stakeholders. Results will additionally be disseminated to the local and research community and the public at large through conference presentations and publication in peer-reviewed journals.